CLINICAL TRIAL: NCT05713994
Title: Combined Hepatic Arterial Infusion Chemotherapy, Tyrosine Kinase Inhibitor/ Anti-VEGF Antibody, and Anti-PD-1/ PD-L1 Antibody as Conversion Therapy for Unresectable Hepatocellular Carcinoma
Brief Title: Combined HAIC, TKI/Anti-VEGF and ICIs as Conversion Therapy for Unresectable Hepatocellular Carcinoma
Acronym: CCGLC-001
Status: Recruiting | Type: Observational
Sponsor: Ze-yang Ding, MD (Other)
Collaborators: Chinese Cooperative Group of Liver Cancer (Other); Chen Xiao-ping Foundation for the Development of Science and Technology of Hubei Province (Other); Haplox Biotechnology Co., Ltd. (Industry); Geneplus-Beijing Co. Ltd. (Industry); The Second Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor-Investigator, Ze-yang Ding, MD, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2020-S205
Record Dates: First submitted 2023-01-16; First posted 2023-02-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Liver Neoplasms; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab; atezolizumab; sintilimab; lenvatinib; Sorafenib; donafenib; regorafenib; apatinib; camrelizumab; Glutamyl Aminopeptidase; spartalizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, urine, and feces. Part of cancer tissue and blood samples are utilized for high-throughput sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- HAIC-A-T cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus bevacizumab (A) and atezolizumab (T) as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Bevacizumab plus Atezolizumab
- HAIC-Len-ICI cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus lenvatinib (Len) and anti-PD-1 antibody as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Lenvatinib; Drug: Anti-PD-1 monoclonal antibody
- HAIC-B-S cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus bevacizumab biosimilar (Byvasda, B) and Sintilimab (Tyvyt, S) antibody as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Bevacizumab Biosimilar IBI305 plus sintilimab
- HAIC-Apa-C cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus Apatinib (Apa) and Camrelizumab (C) antibody as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: apatinib plus camrelizumab
- HAIC-Sor-ICI cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus sorafenib (Sor) and anti-PD-1 antibody as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Sorafenib; Drug: Anti-PD-1 monoclonal antibody
- HAIC-Don-ICI cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus donafenib (Don) and anti-PD-1 antibody as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Donafenib; Drug: Anti-PD-1 monoclonal antibody
- HAIC-Reg-ICI cohort: Patients with advanced hepatocellular carcinoma who was initially evaluated unsuitable for the radical therapy and received combined HAIC plus regorafenib (Reg) and anti-PD-1 antibody as conversion therapy for downstaging.
  Interventions: Procedure: HAIC; Drug: Regorafenib; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Procedure: HAIC — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks.
  Other Names: hepatic arterial infusion chemotherapy of FOLFOX
Drug: Bevacizumab plus Atezolizumab — Bevacizumab (15mg/kg, q3w) plus Atezolizumab (1200 mg, q3w)
  Other Names: Avastin plus Tecentriq
  Groups: HAIC-A-T cohort
Drug: Bevacizumab Biosimilar IBI305 plus sintilimab — Bevacizumab Biosimilar IBI305 (15mg/kg, q3w), and sintilimab (200 mg, q3w)
  Other Names: Byvasda (B) plus S
  Groups: HAIC-B-S cohort
Drug: Lenvatinib — 8mg; p.o.; q.d.
  Other Names: Lenvima
  Groups: HAIC-Len-ICI cohort
Drug: Sorafenib — 400mg; p.o. bid
  Other Names: Nexavar
  Groups: HAIC-Sor-ICI cohort
Drug: Donafenib — 200mg; p.o. bid
  Other Names: Zepsun
  Groups: HAIC-Don-ICI cohort
Drug: Regorafenib — 160 mg; p.o.; q.d.
  Other Names: stivarga
  Groups: HAIC-Reg-ICI cohort
Drug: apatinib plus camrelizumab — Apatinib(250 mg; p.o.; q. d.); camrelizumab (200 mg; iv drip; q2w)
  Other Names: Apa plus C
  Groups: HAIC-Apa-C cohort
Drug: Anti-PD-1 monoclonal antibody — HCC Patients treated with TKI plus anti-PD-1 monoclonal antibody as systemic therapy were recruited. Anti-PD-1 monoclonal antibodies include pembrolizumab (200 mg, q3w), nivolumab (3mg/kg, q2w), camrelizumab (200mg, q2w), tislelizumab (200mg, q3w), sintilimab (200 mg, q3w), or toripalimab (240mg, q3w).
  Other Names: PD-1 inhibitor
  Groups: HAIC-Don-ICI cohort; HAIC-Len-ICI cohort; HAIC-Reg-ICI cohort; HAIC-Sor-ICI cohort

SUMMARY:
This study is conducted to evaluate the efficacy, prognosis, adverse effects, and factors for predicting therapeutic effects and clinical prognosis of combined therapy of hepatic artery infusion chemotherapy (HAIC), tyrosine kinase inhibitor/ anti-VEGF antibody, and anti-PD-1/ PD-L1 antibody for advanced hepatocellular carcinoma which initially unsuitable for the radical therapy, including resection, transplantation, or ablation. Factors are collected in preoperative routine blood examination, preoperative radiological imaging and pathological examination.

DETAILED DESCRIPTION:
As a local interventional treatment, hepatic arterial infusion chemotherapy (HAIC) has shown better efficacy and safety than traditional transcatheter arterial chemoembolization (TACE) in the treatment of unresectable HCC. In addition, HAIC has been widely used as an alternative to sorafenib in advanced HCC in the eastern Asia. Systemic therapies such as tyrosine kinase inhibitors (TKIs), immune checkpoint inhibitors (ICIs), as well as the combined use of anti-VEGF antibody and ICIs have shown promising results in the treatment of advanced HCC. Numerous studies have shown that combination therapy has a trend toward better tumor response rates, survival outcomes, and downstaging rate to monotherapy.

This study is conducted by the by Chinese Collaborative Group of Liver Cancer (CCGLC), the Chinese Chapter of the International Hepato-Pancreato-Biliary Association (CC-IHPBA). It is estimated that 300 patients with advanced hepatocellular carcinoma will be enrolled in about 4 research centers. And it is planned to complete the enrollment within 1 year and it is expected that all enrolled subjects will reach the observation end point in 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Diagnosis of HCC is according to the American Association for the Study of Liver Diseases or European Association for the Study of the Liver guidelines of HCC management;
3. at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or mRESIST criteria;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. Hepatocellular carcinoma (HCC) was assessed as not suitable for radical resection, liver transplant, or ablation treatment after the assessment of a multidisciplinary team because either: (1) R0 resection was not feasible; (2) remnant liver volume was less than 30% in patients who did not have cirrhosis or 40% in patients with cirrhosis, or the results of an indocyanine green test were higher than 15%; (3) patients had Barcelona Clinic Liver Cancer (BCLC) stage B and beyond Up-to-seven criteria; or (4) patients had BCLC stage C.
6. Portal vein involvement (Chen's groups A and B, or Cheng's type I-III) is allowed: Chen's group A1 or Cheng's type I, tumor thrombus is involved in segmental or sectoral branches of the portal vein or above; Chen's group A2 or Cheng's type II, involvement of the first branch of portal vein; Chen's group B or Cheng's type III, involvement of the main portal vein.
7. Hepatic vein invasion (VV1 to VV2) were allowed. Patients with tumor thrombus in inferior vena cava (VV3 type, Sakamoto type 1) can be included; However, patients with inferior vena cava tumor thrombus exceeding the diaphragmatic plane (Sakamoto type II) and reaching the right atrium (Sakamoto type III) cannot be included in the study;
8. Patients with extrahepatic oligometastasis is allowed: extrahepatic oligometastasis was defined as up to three metastatic lesions in up to two organs with the largest diameter of 3 cm
9. Child-Pugh liver function class A-B7
10. No prior transplantation, TACE, or radioembolization to the liver was allowed. Prior locoregional therapies, such as surgical resection, radiotherapy, radiofrequency ablation, percutaneous ethanol injection or cryoablation, are allowed if the disease have progressed since prior treatment. Local therapy must have been completed at least 4 weeks prior to the baseline scan.
11. Adequate organ and marrow function, as defined below:

(1) Hemoglobin≥80 g/L; (2) Absolute neutrophil count ≥1.5 ×10^9/L; (3) Platelet count ≥50 ×10^9/L; (4) Total bilirubin < 51 μmol/L; (5) Alanine transaminase (ALT) and aminotransferase (AST)≤5×ULN; (6) Albumin ≥28 g/L; (7) INR ≤1.6; (8) Serum creatinine < 110 μmol/L.

Exclusion Criteria:

1. Prior invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, lobular or ductal carcinoma in situ of the breast that has been surgically cured
2. Severe, active and uncontrolled co-morbidity including but not limited to:

(1) Persistent or activity (except the HBV and HCV) infection; (2) symptoms of congestive heart failure and uncontrolled diabetes; (3) uncontrolled hypertension, systolic pressure≥160 mmHg or diastolic pressure≥100 mmHg despite anti-hypertension medications≤28 days before randomization or first dose of drug; (4) unstable angina; (5) uncontrolled arrhythmias; (6) active ILD; (7) severe chronic GI disease accompanied by diarrhea; (8) compliance with requirements may limit the research, resulted in significant increase risk of AE or influence Subjects provided psychiatric/social problem status on their ability to provide written informed consent; (9) A history of active primary immunodeficiency or human immunodeficiency virus; (10) Active or previous records of autoimmune disease or inflammatory diseases, including inflammatory bowel disease (e.g., colitis or Crohn's disease], diverticulitis, except [diverticulosis], systemic lupus erythematosus (SLE), sarcoidosis syndrome or Wegener syndrome (e.g., granulomatous vasculitis, gray's disease, rheumatoid arthritis, the pituitary gland inflammation and uveitis]); (11) A history of hepatic decompensation, including refractory ascites, gastrointestinal bleeding, or hepatic encephalopathy.

3. Known to produce allergic or hypersensitive reactions to any study drug or any excipient thereof.

4. Significant clinical gastrointestinal bleeding or a potential risk of bleeding was identified by the investigator during the 30 days prior to study entry.

5. Tumors of the central nervous system, including metastatic brain tumors. 6. Pregnant women or breast-feeding patients. 7. Has received anti-tumor system therapy for HCC. Non-anti-tumor purpose combined hormone therapy (e.g., hormone replacement therapy) is excluded.

8. Is currently using, or has used an immunosuppressive drug within 14 days prior to the first dose of the investigational drug. This standard has the following exceptions: (1) intranasal, inhaled, topical or topical steroids. (e.g., intraarticular); (2) Systemic corticosteroid therapy not exceeding 10 mg/ day of prednisone; (3) prophylactic use of steroids for hypersensitivity. (e.g., CT scan pretherapy medication).

9. A live attenuated vaccine was administered within 30 days prior to the first administration of the study drug. Note: If enrolled, patients shall not receive live attenuated vaccine within 30 days of receiving study drug therapy and after the last administration of study drug.

10. Extrahepatic vascular involvement or thrombosis: superior mesenteric vein (Cheng's type IV), or with inferior vena cava tumor thrombus exceeding the diaphragmatic plane (Sakamoto type II) or reaching the right atrium (Sakamoto type III) cannot be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced hepatocellular carcinoma which initially unsuitable for the radical therapy, including resection, transplantation, or ablation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Amendable to Curative Surgical Interventions | from the date of first treatment to the date of last treatment, an average of 3 years
  Number of patients amendable to curative surgical interventions defined as number of patients receiving curative surgical resection, transplantation, or ablation after successful down-sizing of tumor(s) by intervention.

SECONDARY OUTCOMES:
overall response rate (ORR) measured by mRECIST criteria | rom the date of first treatment to radiographically documented progression according to mRECIST, assessed up to 3 years
  Complete response (CR): Disappearance of any intra-tumoral arterial enhancement in all target lesions; Partial response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Stable disease (SD): Any cases that do not qualify for either partial response or progressive disease; Progressive disease (PD): An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
  ORR=CR+PR.
Time to progression (TTP) | from the date of first treatment to radiographically documented progression according to mRECIST, assessed up to 3 years
  Time to progression (TTP): measured from the date of first treatment to radiographically documented progression according to mRECIST 1.1. This does not include death from any cause.
Time to intrahepatic tumor progression (TTITP) | from the date of first treatment to radiographically documented intrahepatic tumor progression according to mRECIST, assessed up to 3 years
  Time to intrahepatic tumor progression (TTITP): measured from the date of first treatment to radiographically documented intrahepatic tumor progression according to mRECIST 1.1. This does not include death from any cause.
Progression-free survival (PFS) | from the date of first treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 3 years
  measured from the date of first treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Overall survival (OS) | from the date of first treatment to the date of death from any cause, assessed up to 5 years
  Overall survival (OS): measured from date of first treatment to the date of death from any cause. Participants alive or lost to follow-up will be censored at the date of their last visit.
Incidence of Study-Related Adverse Events | from the date of first treatment to 90 days after last treatment, around 3 years and 90 days
  Incidence, nature, and severity of adverse events graded according to the United States National Cancer Institute The Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0)
Pathological response | from the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 5 years
  Pathological response is assessed as the percentage of surface with non-viable cancer cells (represented by necrosis or fibrosis, the ultimate stage of necrosis) in relation to the total tumor area and will be equal to: 100% - viable cancer cells (%). If there are multiple tumors, the mean percentage will be used.
Disease control rate (DCR) | from the date of first treatment to radiographically documented response according to mRECIST, assessed up to 3 years
  Percentage of patients that had a CR, PR, or SD ≥ 6 months per mRECIST
Duration of response | from the date of first documented evidence of CR or PR to first documented sign of PD or death from any cause according to mRECIST 1.1, assessed up to 3 years
  Defined as the time from first documented evidence of CR or PR until the first documented sign of disease progression (PD) or death from any cause
Quality of Life (QoL) after treatment | assessed form the date of first followup to radiographically documented progression or or death from any cause, up to 3 years
  The life quality of every subject is assessed every 3 months during follow up according to the 45-item FACT-Hep questionnaire, which assesses generic HRQL concerns and disease-specific issues.

CONTACTS AND LOCATIONS:
Overall Officials: Wanguang Zhang, M.D., Study Chair — Tongji Hospital
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - TongjiHospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazzaferro V, Citterio D, Bhoori S, Bongini M, Miceli R, De Carlis L, Colledan M, Salizzoni M, Romagnoli R, Antonelli B, Vivarelli M, Tisone G, Rossi M, Gruttadauria S, Di Sandro S, De Carlis R, Luca MG, De Giorgio M, Mirabella S, Belli L, Fagiuoli S, Martini S, Iavarone M, Svegliati Baroni G, Angelico M, Ginanni Corradini S, Volpes R, Mariani L, Regalia E, Flores M, Droz Dit Busset M, Sposito C. Liver transplantation in hepatocellular carcinoma after tumour downstaging (XXL): a randomised, controlled, phase 2b/3 trial. Lancet Oncol. 2020 Jul;21(7):947-956. doi: 10.1016/S1470-2045(20)30224-2. PMID 32615109
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160